CLINICAL TRIAL: NCT05593133
Title: Comparative Effects of PNF and Gait Training Exercises on Balance and Gait in Patients With Diabetic Neuropathy
Brief Title: PNF and Gait Training on Balance and Gait in Diabetic Neueopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maryam Rauf
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Neuropathies
Keywords: PNF; DGI; BBS; TAT; MNSI
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pnf exercises (Experimental): warm up, rhythmic stabilization, hold relax, contract relax and light exercises performed on three muscle groups
  Interventions: Other: Pnf exercises
- Gait training exercises (Experimental): exercises comprised of one foot balancing, leg raises, heel raises, tight-rope walking.
  Interventions: Other: Gait training exercises

INTERVENTIONS:
Other: Pnf exercises — PNF techniques will comprise of Warm up, Rhythmic stabilization, Hold Relax, Contract Relax and light exercises and performed on three muscle groups ( Hamstring, Quad and Calf).
  20 participants will be followed up with the therapist regularly twice a week for 30 minutes session each for a duration of 8 weeks.
  Arms: Pnf exercises
Other: Gait training exercises — gait Training exercises comprised of one foot balancing, leg raises, heel raises, tight-rope walking. 20 participants will be followed up with the therapist regularly twice a week for 30 minutes session each for a duration of 8 weeks.
  Arms: Gait training exercises

SUMMARY:
To determine the effects of PNF and Gait Training Exercises on Balance and Gait in diabetic neuropathy patients . 40 patients will be explained in detail about the study procedure. Informed consent will be taken. Patients will be divided in two groups each consisting of 20 people.

Subjects will be evaluated using the Michigan Neuropathy Screening Questionnaire (screening tool) . One group will be tested by PNF techniques and the second group will be tested by Gait Training exercises.

Balance will be assessed by Berg Balance scale (BBS) and Tinetti scale before, during and after the study to assess risk of fall and injury. Gait will be assessed by Dynamic Gait index in the same manner. All patients will be followed up with the therapist regularly twice a week for 30 minutes session each for a duration of 8 weeks.

DETAILED DESCRIPTION:
Objective To determine the effects of PNF and Gait Training Exercises on Balance and Gait in diabetic neuropathy patients Hypothesis Null hypothesis : There is no difference between PNF and Gait Training Exercises.

Alternative hypothesis : There is difference between PNF and Gait Training Exercises

Methodology (Design, sample size, sampling technique, inclusion and exclusion criteria and tool) Study design: This study is Randomized Clinical Trial Sample size: Sample size will be 40 (Two groups of 20 each) Assumed standard deviation=6.5 Confidence interval= 0.95 Desired precision=2 Calculated by epitool. Sampling technique: Convenient sampling will be used to collect data. Study design setting: Data will be conducted from Hospital wards and Outpatient departments

Inclusion Criteria:

Both male and female in the age group Patients suffering from Diabetes Mellitus (Type 1, Type 2), suffering From effects of diabetic neuropathy such as Gait instability, imbalance, numbness, tingling, Paresthesia in lower limbs for a duration of at least three months.

* HbA1c more than 7 from 6 months.
* Score higher than 7 out of 15 in the Michigan Neuropathy questionnaire scale and Examination score higher than 2.5.

Exclusion Criteria:

* Patients suffering from significant CNS dysfunctions.
* Musculoskeletal deformities
* Vestibular dysfunction
* Internal ear infections
* Complete sensory loss
* Hypoglycemia
* Lower extremity arthritis or pain that limits standing or weight bearing. Data collection procedure All 40 patients will be explained in detail about the study procedure. Informed consent will be taken. Patients will be divided in two groups each consisting of 20 people.

Subjects will be evaluated using the Michigan Neuropathy Screening Questionnaire (screening tool) . One group will be tested by PNF techniques and the second group will be tested by Gait Training exercises.

PNF techniques will comprise of Warm up, Rhythmic stabilization, Hold Relax, Contract Relax and light exercises and performed on three muscle groups ( Hamstring, Quad and Calf).

Gait Training exercises will comprise of One Foot Balancing, Leg raises, Heel raises, Tight-rope Walking.

Balance will be assessed by Berg Balance scale (BBS) and Tinetti scale before, during and after the study to assess risk of fall and injury. Gait will be assessed by Dynamic Gait index in the same manner. All patients will be followed up with the therapist regularly twice a week for 30 minutes session each for a duration of 8 weeks.

ELIGIBILITY:
Inclusion criteria:

Both male and female in the age group 40-65 • Patients suffering from Diabetes Mellitus (Type 1, Type 2), suffering From effects of diabetic neuropathy such as Gait instability, imbalance, numbness, tingling, Paresthesia in lower limbs for a duration of at least three months.

* HbA1c more than 7 from 6 months.
* Score higher than 7 out of 15 in the Michigan Neuropathy questionnaire scale and Examination score higher than 2.5.

Exclusion Criteria:

* Patients suffering from significant CNS dysfunctions.

  * Musculoskeletal deformities
  * Vestibular dysfunction
  * Internal ear infections
  * Complete sensory loss

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
tinnete scale | 8 weeks
  The test requires a hard armless chair, a stopwatch and also, a 15 feet even and uniform walkway. It has 2 sections: one assesses balance abilities in a chair and also in standing; the other assesses dynamic balance during gait on a 15 feet even walkway.Next, the patient will have to walk a few meters at a normal speed, followed by turning and walking back at a "fast but safe" speed. The patient will then sit back down. As well as in the first part of the test, there are some points the evaluator has to look at. These are the length and height of the steps, the symmetry and continuity of the steps and straightness of the trunk.
  During this test, the patient can use any assistive devices (walking stick, crutches, zimmer frame) they would normally use
Berg Balance Scale | 8 weeks
  Document each task and/or give instructions as written. When scoring, please record the lowest response category that applies for each item.
  In most items, the subject is asked to maintain a given position for a specific time. Progressively more points are deducted if:
  the time or distance requirements are not met the subject's performance warrants supervision the subject touches an external support or receives assistance from the examiner The subject should understand that they must maintain their balance while attempting the tasks. The choices of which leg to stand on or how far to reach are left to the subject. Poor judgment will adversely influence the performance and the scoring.
  Equipment required for testing is a stopwatch or watch with a second hand, and a ruler or other indicator of 2, 5, and 10 inches. Chairs used during testing should be a reasonable height. Either a step or a stool of average step height may be used for item.
Dynamic Gait index | 8 weeks
  8 functional walking tests are performed by the subject and marked out of three according to the lowest category which applies. 24 is the total individual score possible. Scores of 19 or less have been related to increase incidence of falls.
  Equipment needed
  Box (Shoebox), Cones (2), Stairs, 20' walkway, 15" wide
  Completion Time
  15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Azam, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Central Park Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No